CLINICAL TRIAL: NCT06373328
Title: Post-Pandemic Genomic Epidemiology of Pneumococcal Carriage Among Children and Adults in the General US Population
Brief Title: Post Pandemic Pneumococcal Carriage Among Children and Adults
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: Merck Sharp & Dohme Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00006081
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pneumococcal Carriage
Keywords: Nasopharyngeal; Children; Pandemic; Genomic; Epidemiology; Pneumococcal Carriage; Streptococcus pneumoniae

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biospecimens from participants of the study will be coded and de-identified by the clinical research coordinators and will be accompanied by corresponding clinical data collected at the time of biospecimen collection. De-identified biospecimens will be stored at -80°C indefinitely.
  Data received with the biospecimens and from the analyses generated in the study will be stored electronically on a dedicated password protected server at the Burnett School of Biomedical Sciences and accessed only through UCF computers. Access to this data will be limited to the research personnel involved in the analyses.
  Biospecimens will be accessed only by authorized personnel working in the PIs laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children: This is a non-interventional study with data collection online, chart review, and biospecimen collection (nasopharyngeal swab). The swab will then be used for biomarker discovery.
  Findings will be compared and analyzed between the children and adult groups.
- Adults: This is a non-interventional study with data collection online, chart review, and biospecimen collection (nasopharyngeal swab). The swab will then be used for biomarker discovery.
  Findings will be compared and analyzed between the children and adult groups.

SUMMARY:
The PI propose to conduct a genomic epidemiology study of pneumococcal carriage among children and adults in a large metropolitan city. These data will allow PI to assess the post-pandemic population structure, investigate the phylogenetic relationship between isolates from children and adults, and compare pneumococcal populations across diverse geographic areas.

DETAILED DESCRIPTION:
The SARS-CoV-2 pandemic profoundly impacted human health directly and indirectly. As such, elucidating pre- and post-pandemic trends in the epidemiology and population genomics of human respiratory pathogens including those such as the bacteria Streptococcus pneumoniae, a human commensal and the causative agent of invasive pneumococcal disease (IPD), merits study.

Nasopharyngeal samples will be processed at the PIs Laboratory to identify S. pneumoniae. If present, the isolate will undergo bacterial whole genome sequencings and population dynamic analysis. Carriage prevalence and serotype composition will be compared to extant studies and pneumococcal genomic data will be analyzed in the context of samples from the US and abroad.

ELIGIBILITY:
Inclusion Criteria:

* Children, ages 7 to 59 months (less than 5 years)
* Adults, ages 50 and older
* Ability to provide informed consent (from parents for children participants)
* ability to read and speak in English
* Agree to comply with study procedures (complete online data questionnaire and provide a nasopharyngeal collection).

Exclusion Criteria:

* Have been on an antibiotic in the last 2 weeks
* Have a respiratory infection that would make an nasopharyngeal collection improbable
* Have underlying developmental or chronic conditions impacting immune or respiratory function (e.g., immunocompromised, cystic fibrosis, cerebral palsy, paralysis)
* Adults unable to consent, individuals who are not yet adults, and prisoners will be excluded from this study.

Min Age: 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The PI seeks to recruit 450 children 7-59 months of age and 450 adults 50 years or older over a 16-month period. Children will be equally distributed between 7-23 months and 24-59 months and adults equally distributed in the age ranges: 50-64 years, 65-74 years, and 75 years or older.
  Pregnant women may choose to be in the study. The study procedures do not pose a risk to the safety of the unborn child or the woman.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pneumococcal carriage prevalence and distribution of serotypes among children and adults calculated from the results of S. pneumoniae isolation using qPCR. | 22 months

SECONDARY OUTCOMES:
Phylogenetic relationship of pneumococcal isolates collected among child and adult populations using whole-genome sequencing libraries. | 22 months
Putative transmission networks between children and adult populations from online questionnaires. | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Taj Azarian, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No